CLINICAL TRIAL: NCT05610449
Title: Assessing Performance of the Testing Done Simple Covid 19 Antigen Test
Status: Completed | Type: Observational
Sponsor: Testing Done Simple (Industry)
Collaborators: Nao Medical Urgent Care (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7113211
Record Dates: First submitted 2022-11-07; First posted 2022-11-09 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Antigen test; Test; Diagnosis
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Testing Done Simple Antigen test in Symptomatic Subjects (Nasal swab)
  Interventions: Diagnostic Test: Testing Done Simple SARS CoV-2 Antigen Test
- Testing Done Simple Antigen test in Asymptomatic Subjects (Nasal swab)
  Interventions: Diagnostic Test: Testing Done Simple SARS CoV-2 Antigen Test

INTERVENTIONS:
Diagnostic Test: Testing Done Simple SARS CoV-2 Antigen Test — Collections of specimens from subjects presenting with Covid-19 like symptoms or known/suspected exposure to SARS CoV-2 via nasal swabs administered by trained medical personnel.

SUMMARY:
This study will measure the sensitivity and specificity of the Testing Done Simple severe acute respiratory syndrome (SARS) CoV-2 antigen test in subjects with suspected Covid-19 that present throughout several urgent care clinics. The antigen test performance will be compared to a real-time polymerase chain reaction (RT-PCR) test.

DETAILED DESCRIPTION:
The Testing Done Simple antigen test is a lateral flow immunoassay that detects the presence of the SARS CoV-2 nucleoprotein and is primarily intended for use in an at home setting. The antigen test will be compared to a traditional RT-PCR tested nasal swab specimens. The purpose of study is to measure the performance of the Testing Done Simple test via sensitivity and specificity when compared to the gold-standard RT-PCR test. The test will be administered in symptomatic and asymptomatic subjects and participants will report the days that has passed since their symptom onset. The RT-PCR test will be performed prior to the Testing Done Simple test.

ELIGIBILITY:
Inclusion Criteria:

* Subject was given a SARS CoV 2 PCR test for any of the following 4 reasons:

  1. Subject has Covid like symptoms that started within past (7) days
  2. Subject has been exposed to another individual with a known Covid diagnosis or probable Covid diagnosis
  3. Subject needs Covid test done for travel, school, work, etc
  4. Subject works in a high risk environment
* Subject can provide a nasal swab sample
* Subject is at least 18 years of age
* Subject was given a SARS CoV 2 PCR test on same day participating this study
* Subject provides informed consent

Exclusion Criteria:

* Subject is less than 18 years of age
* Subject does not provide consent
* Subject's Covid 19 related symptom(s) started greater than 7 days from visit
* Asymptomatic subjects whom have had symptom(s) within past (14) days
* Signs of local infection in the area of the face
* Subject was not given a SARS CoV 2 PCR test on same day as study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohorts consist of a symptomatic group of patients with Covid related symptoms and an asymptomatic group of patients that may have been exposed to Covid through another person
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 15 minutes
  Sensitivity (True Positive Rate) of Testing Done Simple Antigen Test compared to RT-PCR
Specificity | 15 minutes
  Specificity (True Negative Rate) of Testing Done Simple Antigen Test compared to RT-PCR

SECONDARY OUTCOMES:
Sensitivity in Relation to the Time Since Symptom Onset in Symptomatic subjects | 15 minutes
  Sensitivity of Testing Done Simple Antigen Test according to the days of symptom onset in symptomatic subjects

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nao Medical Urgent Care-Astoria, Queens, New York
  - Nao Medical Urgent Care-Jackson Heights, Queens, New York

IPD SHARING:
Plan to Share IPD: No